CLINICAL TRIAL: NCT06123000
Title: Modified Widman Flap (MWF) vs Fibre Retention Osseous Resective Surgery (FibReORS): A Randomized, Controlled, Clinical Trial.
Brief Title: Modified Widman Flap vs Fibre Retention Osseous Resective Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Luigi Barbato, Principal Investigator, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MWF vs FibReORS
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis; Periodontal Pocket; Periodontal Attachment Loss
MeSH Terms: conditions — Periodontitis; Periodontal Pocket; Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Widman Flap (MWF) (Active Comparator): At buccal and lingual/palatal side, a full thickness incision parallel to the long axis of the tooth will be performed. In case of buccal or lingual pockets deeper than 2 mm, this initial incision will be placed approximately 1 mm apically to the free gingival margin. All soft tissues will be removed from the bony surface of intrabony defects. In case of incomplete adaptation between the flaps and the teeth or between the buccal and lingual flaps, the flaps will be thinned, and an amount of bone removal will be performed. Only osteoplasty will be allowed, while these patients will not receive ostectomy.
  Interventions: Procedure: Modified Widman Flap (MWF)
- Fiber Retention Osseous Resective Surgery (FibReORS) (Experimental): At the buccal sites, internally beveled incisions will be positioned at intra-sulcular or extra-sulcular level based on the apico-coronal dimension of the keratinized tissue. A split thickness flap beyond the MGJ will be then elevated. Vertical releasing incisions will be used to augment surgical access as needed. At lingual site split-full-thickness flap was used positioning an extra-sulcular internally beveled primary incision, while at the palatal area, the thinned palatal flap technique will be performed
  Interventions: Procedure: Fiber Retention Osseous Resective Surgery (FibReORS)

INTERVENTIONS:
Procedure: Modified Widman Flap (MWF) — At buccal and lingual/palatal side, a full thickness incision parallel to the long axis of the tooth will be performed. In case of buccal or lingual pockets deeper than 2 mm, this initial incision will be placed approximately 1 mm apically to the free gingival margin. All soft tissues will be removed from the bony surface of intrabony defects. In case of incomplete adaptation between the flaps and the teeth or between the buccal and lingual flaps, the flaps will be thinned, and an amount of bone removal will be performed. Only osteoplasty will be allowed, while these patients will not receive ostectomy.
  Arms: Modified Widman Flap (MWF)
Procedure: Fiber Retention Osseous Resective Surgery (FibReORS) — At the buccal sites, internally beveled incisions will be positioned at intra-sulcular or extra-sulcular level based on the apico-coronal dimension of the keratinized tissue. A split thickness flap beyond the MGJ will be then elevated. Vertical releasing incisions will be used to augment surgical access as needed. At lingual site split-full-thickness flap was used positioning an extra-sulcular internally beveled primary incision, while at the palatal area, the thinned palatal flap technique will be performed.
  Arms: Fiber Retention Osseous Resective Surgery (FibReORS)

SUMMARY:
The treatment of periodontitis should be carried out in an incremental manner, first by achieving adequate patient's oral hygiene practices and risk factor control during the first step of therapy and then, during the second step of therapy, by professional elimination (reduction) of supra and subgingival biofilm and calculus.

If the endpoints of therapy (no periodontal pockets >4 mm with bleeding on probing, BoP, or deep pockets ≥5 mm) have not been achieved, the third step of therapy should be implemented.

In fact, residual pockets following step 1 and 2 of periodontal treatment are associated with increased risk of periodontal disease progression in the long-term as reported by Claffey & Egelberg in1995. Residual probing depth (PPD) ≥5 mm after active therapy is a risk factor for disease progression and tooth loss during supportive periodontal therapy (SPT), suggesting that additional treatment of residual pockets is strongly recommended.

The third step of treatment includes the following interventions: repeated subgingival instrumentation, access flap periodontal surgery, resective periodontal surgery, regenerative periodontal surgery.

In case of residual pockets associated with shallow-moderate infrabony defects at posterior teeth, where both regenerative therapy and non-surgical re-instrumentation are usually not indicated, access flap procedures (i.e., the Modified Widman Flap, MWF) and the Osseous Resective Surgery (ORS) are considered two of the most viable options.

The value of these surgical techniques has been tested over the years by different clinical trials, and the choice of a surgical approach still relies mainly on the decision-making process of the surgeon, since the long-term outcomes of the different periodontal surgical procedures are similar, as highlighted by a recent systematic review.

Nevertheless, one the main criticism that have been moved against ORS, lies on the fact that the side effects (i.e., gingival recessions) seem to be more severe for ORS surgery, when compared with MWF.

In the early 2000s, Carnevale proposed the Fibre Retention Osseous Resective Surgery (FibReORS), an approach that leads to a more conservative bone resection to eliminate infrabony defects and establish a positive bony architecture than the conventional ORS. Indeed, this one, based on the histological findings by Gargiulo et al. (1961), uses the level of the connective tissue attachment - rather than the bottom of the osseous defect - as the reference to apply the principles of ORS.

Two randomized clinical trials demonstrated that FibReORS is similarly effective as ORS for PPD reduction with less final gingival recessions (REC), clinical attachment loss (CAL) patient morbidity.

Nevertheless, no studies have ever directly compared FibreORS with MWF. Therefore, the aim of this randomized clinical trial (RCT) is to compare the efficacy of FibReORS versus MWF in the treatment of periodontal pockets associated with infrabony defects ≤3 mm at posterior natural teeth.

Objectives

The experimental hypothesis is:

FibReORS is superior to MWF in achieving PPD closure (PPD <4 mm without BoP) at posterior teeth associated with shallow-moderate infrabony defects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients affected by periodontitis;
* No systemic disease or pregnancy;
* No systemic antibiotic therapy in 6 months preceding the enrollment;
* Smoking ≤ 20 cigarettes/day;
* Full-mouth plaque score (FMPS) and full- mouth bleeding score (FMBS) ≤ 15%;
* Residual periodontal pocket ≥5 mm with bleeding on probing at posterior natural teeth;
* Experimental pocket associated with a detectable infrabony defect ≤ 3mm at x-ray;
* No history of periodontal surgery at the experimental site.

Exclusion Criteria:

* Undetectable cemento-enamel junction (CEJ) at experimental teeth;
* Severe furcation involvement (class II and III);
* Abutment for prosthetic rehabilitation;
* Periodontal Pockets associated with infrabony defect >3 mm;
* Horizontal bone loss higher than 1/3 of the root length at experimental teeth;
* Severe tooth mobility at baseline (class 2 or 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Periodontal Pocket Closure | Six months after the procedure
  Distance between the tip of a periodontal probe and the gingival margin < 4 mm, without bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No